CLINICAL TRIAL: NCT00005224
Title: Gender Response To Coronary Risk
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1103; R01HL040368 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine sex differences in behavioral and psychosocial variables such as occupation, Type A behavior, and hostility as they related to primary coronary risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Although coronary heart disease is a major factor in morbidity and mortality in both sexes, most studies prior to 1988 when the study was initiated focused on men and overlooked the magnitude of the problem in women. Coronary heart disease mortality and morbidity rates are higher in men than in women, accounting for 41 percent of the sex difference in overall mortality in the United States. Women's advantage, however, does not seem to be stable over time nor universal. For example, in 1920, the age adjusted ratio of male to female coronary heart disease deaths was approximately equal, but between 1975 and 1978, it has increased to a level of 2.47 in the United States. Also, sex mortality ratios for heart disease differ widely across countries ranging from 5/1 in Finland to 1.87/1 in Yugoslavia. Thus, relying on biological differences alone when explaining this sex differential is not convincing.

Based on Framingham data, among the most important risk factors predicting coronary heart disease in both women and men are--aside from age--cholesterol, cigarette smoking, and blood pressure. Consistent with the observation that men are more likely to fall victim to coronary heart disease than women is the fact that they also exhibit higher levels of these risk factors when compared to women, at least up to the age of 45. Standardization of risk factor levels and controlling for both levels of risk factors on coronary heart disease probabilities eliminated the sex differential in 45 to 54 year olds of the Framingham Study. However, among the 55 to 74 year olds, the sex differential was not due to differences in levels or impact of the risk factors. It was conceivable that the sex mortality differential at the older ages was due to the sex differential in primary coronary risk factors at the younger ages.

Of particular interest was the fact that the primary risk factors appeared to be influenced by behavior. It was possible that gender differences in behavior might explain gender differences in primary coronary risk factors. Alternatively, there was some evidence that the primary coronary risk factors were not solely responsible for the etiology of coronary heart disease. Gender differences in psychosocial variables, such as Type A behavior, hostility, and occupational stress that might play independent roles in the etiology of coronary heart disease had not been systematically investigated.

DESIGN NARRATIVE:

Gender differences in primary risk factors were determined, with all analyses being controlled for body mass since men score higher on body mass index than women and body mass is related to levels of primary coronary risk factors. One-way analyses of covariance were performed for plasma lipids and lipoproteins, blood pressure, and heart rate. Gender differences in psychosocial variables associated with coronary risk were investigated. Analyses were performed on primary coronary risk factors at baseline in order to investigate the relationships of occupational characteristics such as demand and control with age and body mass index. Covariance analyses were performed for Type A/Type B by high and low occupational control and by high and low demand for each sex. The role of parental history of heart disease, Type A behavior and smoking in elevated primary coronary risk factors among oral contraceptive users were also investigated.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1990-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerdi Weidner — State University of New York

REFERENCES:
- [Background] Weidner G, Friend R, Ficarrotto TJ, Mendell NR. Hostility and cardiovascular reactivity to stress in women and men. Psychosom Med. 1989 Jan-Feb;51(1):36-45. doi: 10.1097/00006842-198901000-00004. PMID 2928459
- [Background] Emmons KM, Weidner G, Collins RL. Smoking cessation and cardiovascular reactivity to stress. J Behav Med. 1989 Dec;12(6):587-98. doi: 10.1007/BF00844827. PMID 2634111
- [Background] Weidner G, Helmig L. Cardiovascular stress reactivity and mood during the menstrual cycle. Women Health. 1990;16(3-4):5-21. doi: 10.1300/J013v16n03_02. PMID 2267809
- [Background] Weidner G, Connor SL, Chesney MA, Burns JW, Connor WE, Matarazzo JD, Mendell NR. Sex differences in high density lipoprotein cholesterol among low-level alcohol consumers. Circulation. 1991 Jan;83(1):176-80. doi: 10.1161/01.cir.83.1.176. PMID 1984880
- [Background] Hutt J, Weidner G. The effects of task demand and decision latitude on cardiovascular reactivity to stress. Behav Med. 1993 Winter;18(4):181-8. doi: 10.1080/08964289.1993.9939113. PMID 8461490
- [Background] Weidner G, Connor SL, Hollis JF, Connor WE. Improvements in hostility and depression in relation to dietary change and cholesterol lowering. The Family Heart Study. Ann Intern Med. 1992 Nov 15;117(10):820-3. doi: 10.7326/0003-4819-117-10-820. PMID 1416556
- [Background] Emmons KM, Weidner G, Foster WM, Collins RL. Improvement in pulmonary function following smoking cessation. Addict Behav. 1992;17(4):301-6. doi: 10.1016/0306-4603(92)90036-u. PMID 1502964
- [Background] Weidner G, Hutt J, Connor SL, Mendell NR. Family stress and coronary risk in children. Psychosom Med. 1992 Jul-Aug;54(4):471-9. doi: 10.1097/00006842-199207000-00009. PMID 1502288